CLINICAL TRIAL: NCT00190814
Title: Efficacy and Safety of Duloxetine Compared With Placebo in Women With Symptoms of Mixed Urinary Incontinence.
Brief Title: Effectiveness and Safety of Duloxetine in Women Experiencing Urinary Leakage Due to Physical Stress and Urge.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6192; F1J-MC-SBBO
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Urinary Incontinence, Stress
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: duloxetine
Drug: placebo

SUMMARY:
The purpose of the study is to evaluate the effectiveness of duloxetine in reducing urinary incontinence(leakage of urine)occurrences in women due to physical stress and leakage that occurs during a strong need(urge) to urinate.

ELIGIBILITY:
Inclusion Criteria:

* female outpatients greater than or equal to 18 years of age.
* experience episodes of urinary incontinence based on diagnostic criteria of at least 4 episodes a week with symptoms for a minimum of three months prior to start of study.
* have an educational level and degree of understanding English.
* are free of urinary tract infections.
* have a discreet episodes of incontinence(i.e. dry between episodes and do not continuously leak.)

Exclusion Criteria:

* have received treatment for incontinence within the last 5 years.
* suffer from severe constipation.
* currently nursing or breast feeding.
* any nervous system disease that would affect normal urinary function.
* any extension of internal organs beyond the vaginal opening.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2003-09; Study Completion 2006-05

PRIMARY OUTCOMES:
The study purpose is to assess the efficacy of duloxetine 40 mg BID for up to 8 weeks in women with mixed urinary incontinence(MUI) compared with placebo as measured by: the change in total incontinence episode frequency(IEF) from baseline to endpoint.

SECONDARY OUTCOMES:
Additional assessments of incontinence episode frequency using various standardized instruments will be performed.
To monitor the safety of duloxetine based on clinical laboratory values and the occurrence of treatment-emergent adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559) Monday-Friday 9am-5pm Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY(1-877-285-4559, 1-317-615-4559), Monday-Friday, 9 am to 5 pm Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Baltimore, Maryland, United States
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY(1-877-285-4559, 1-317-615-4559), Monday-Friday, 9 am to 5 pm Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, London, Ontario, Canada
- For additional information regarding investigative sites for this trial, please call 1-877-CTLILLY(1-877-285-4559, 1-317-615-4559), Monday-Friday, 9 am to 5 pm Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, London, United Kingdom